CLINICAL TRIAL: NCT06706232
Title: Acceptability & Safety of Two Sequential Doses of Psilocybin in Bipolar Disorder II Depression and Suicidality
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Anne and Don Fizer Foundation (Unknown)
Responsible Party: Principal Investigator, Thomas D. Meyer, PhD, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0905
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Bipolar II Disorder; Depression, Bipolar; Suicidality
Keywords: Bipolar II Depression; Psilocybin
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation | interventions — Psilocybin; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin with therapeutic support (Experimental): Up to two sequential administrations of 25 mg psilocybin with additional therapeutic support.
  Interventions: Drug: Psilocybin; Behavioral: Therapeutic Support

INTERVENTIONS:
Drug: Psilocybin — Two sequential administrations of 25 mg psilocybin, 4 weeks apart.
Behavioral: Therapeutic Support — Five preparatory in-person psychotherapy sessions will be offered before the first administration session during weeks 1, 2, 3, 4, and 5. The optional second administration session will be preceded by a shorter 60 min preparatory session the day before.
  Each administration session will be followed by 3 integration sessions and will adopt a Mindfulness-based CBT approach (M-CBT), in which a therapist will help the participant to process their experience and how to translate this into actual changes in everyday life.
  If participants prefer more psychological support after the second administration session, they will be offered additional, optional therapy sessions for the duration of the trial regardless if they opted for a second administration session or not.

SUMMARY:
The purpose of the study is to assess the safety and acceptability of up to two sequential administrations of 25 mg psilocybin with additional therapeutic support in decreasing suicidality in patients with Bipolar Disorder (BD II) depression.

DETAILED DESCRIPTION:
This study aims to determine whether psilocybin paired with psychotherapy is a safe, feasible, and acceptable treatment for Bipolar II (BD II) depression, specifically, individuals experiencing suicidal ideation (without having an active plan or intention to act). The design is a non-randomized clinical trial, where patients will receive up to 2 doses of 25mg psilocybin in the context of psychological support informed by mindfulness-based CBT and typical elements of psychedelic treatments (e.g., preparation, intention setting, integration). The investigators will measure suicidality, depression, and acute experiences using validated questionnaires at multiple time points in the study. If this study shows psilocybin to be a feasible, acceptable, and safe treatment option, this would have huge implications for improving outcomes because highly effective treatment for suicidality in patients with Bipolar Disorder is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed written informed consent
* Must be at 25 years of age or older at screening (but below age of 70)
* Confirmed Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of BD-II using clinical records and Diagnostic Interview for Anxiety, Mood, and Obsessive-compulsive disorder (OCD) and Related Neuropsychiatric Disorders (DIAMOND)
* Must meet criteria for suicidality according to the INQ cutoff scores: A score of at least 12 on the Perceived Burden (PB) subscale and at least a score of 36 on the Thwarted Belongingness (TB) subscale indicating substantial risk for passive suicidal ideation
* Must meet criteria for depression according to the MADRS cutoff scores: A score of 7-34 indicating mild to moderate depression
* Must pass medical examination (physical exam, personal/family medical history, including consultation with current medical provider, ECG, about 4 tablespoons blood draw, psychiatric/psychological assessments, urine drug test)
* Willingness to taper down mood stabilizers and other relevant medications (including but not limited to: antidepressants, antipsychotics, lithium, benzodiazepines, Monoamine oxidase inhibitors (MAOIs), Selective serotonin reuptake inhibitors (SSRIs), Serotonin and norepinephrine reuptake inhibitors (SNRIs), A serotonin-norepinephrine-dopamine reuptake inhibitors (SNDRIs), Tricyclic antidepressants (TCAs), stimulants, cannabis, and other medications, supplements or therapeutics that affect serotonergic function) for the duration of the study before and during administration days (starting 5 weeks before administration), and be off medication for at least 2 weeks prior to administration
* Willingness to stop allowed medication at least 24 h prior to administration of psilocybin as advised by study physician (e.g., benzodiazepines)
* Ability to complete all protocol required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits

Exclusion Criteria:

* Participants who do not read/speak English
* Active suicidal ideation with at least some intent and/or plan (i.e., a current score of 4 or 5 on the C-SSRS)
* History of medically significant suicide attempt in the last 6 months
* Current or past history of Bipolar I disorder, psychotic symptoms or psychotic disorder, (including but not limited to schizophrenia, delusional disorder, schizoaffective disorder) clinically relevant personality disorder (such as borderline, antisocial, narcissistic or paranoid personality disorder), or any serious psychiatric comorbidity considered negatively impacting participation or safety (e.g., PTSD or severe substance use or alcohol disorder) assessed by medical history and/or a structured clinical interview
* Have a first or second degree relative with Bipolar I disorder or a psychotic disorder
* Currently experiencing a hypomanic or mixed-symptom episode
* Have a psychiatric or other condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* Any indication of a Personality Disorder (PD) such as but not limited to Borderline, Narcissistic, Antisocial, Paranoid, or Schizotypal PD based on Structured Clinical Interview for DSM-5 for PD and/or clinical judgment

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility as Assessed by Number of Participants who Complete the Trial (Overall Retention) | from baseline to 3 weeks after first administration session
  This is assessed by number of participants who complete the trial, that is, the number of participants who complete the first dose and follow-up visits up to 3 weeks after the first dose.
Feasibility as Assessed by Number of Therapy Sessions Attended | from baseline to 3 weeks after first administration session
Feasibility as Assessed by Number of Assessments Completed | from baseline to 3 weeks after first administration session
Acceptability of Two Dosing Sessions as Assessed by Number of Participants who Choose to Participate in a Second Administration Session | 11 weeks after first administration session
Acceptability as Assessed by Number of Therapy Sessions Attended | from baseline to 11 weeks after first administration session
Acceptability as Assessed by Number of Assessments Completed | from baseline to 11 weeks after first administration session
Score on the Thwarted Belongingness (TB) Items of the Interpersonal Needs Questionnaire (INQ-15) | baseline, 3 weeks after first administration session
  The Thwarted Belongingness (TB) section of the INQ-15 has a total score range from 9 to 63, with a higher score indicating greater TB.
Score on the Perceived Burdensomeness (PB) Items of the Interpersonal Needs Questionnaire (INQ-15) | baseline, 3 weeks after first administration session
  The Perceived Burdensomeness (PB) section of the INQ-15 has a total score range from 6 to 42, with a higher score indicating greater PB.
Score on the Columbia-Suicide Severity Rating Scale (C-SSRS) | baseline, 3 weeks after first administration session
  The total score on the C-SSRS ranges from 0-5, with 5 indicating the highest level of suicidal ideation.

SECONDARY OUTCOMES:
Score on the Montgomery-Åsberg Depression Rating Scale (MADRS) | baseline, 3 weeks after first administration session
  The total score on the MADRS ranges from 0 to 60, with a higher score indicating a greater depression.
Score on the Quick Inventory of Depressive Symptomatology (QIDS-SR16) | baseline, 3 weeks after first administration session
  Total score on the QIDS-SR16 ranges from 0 to 27, where higher scores indicate a higher occurence of depressive symptoms.
Score on the Young Mania Rating Scale (YMRS) | baseline, 3 weeks after first administration session
  The total score on the YMRS ranges from 0 to 60, with higher scores indicating greater severity of mania.
Psychiatric Symptoms as Assessed by Score on the Brief Psychiatric Rating Scale (positive symptom subscale) (BPRS+) | baseline, 3 weeks after first administration session
  The total score on the BPRS+ ranges from 4 to 28, with higher scores indicating a higher severity of psychopathology.
Score on the Altman Self-Rating Mania Scale (ASRM) | baseline, 3 weeks after first administration session
  The total score on the ASRM ranges from 5-25, with higher scores indicating more severity of mania.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson ST, van der Vaart A, Miller T, LaPratt J, Swartz K, Shoultz A, Lauterbach M, Sackeim HA, Suppes T. Single-Dose Synthetic Psilocybin With Psychotherapy for Treatment-Resistant Bipolar Type II Major Depressive Episodes: A Nonrandomized Open-Label Trial. JAMA Psychiatry. 2024 Jun 1;81(6):555-562. doi: 10.1001/jamapsychiatry.2023.4685. PMID 38055270
- [Background] Bogenschutz MP, Ross S, Bhatt S, Baron T, Forcehimes AA, Laska E, Mennenga SE, O'Donnell K, Owens LT, Podrebarac S, Rotrosen J, Tonigan JS, Worth L. Percentage of Heavy Drinking Days Following Psilocybin-Assisted Psychotherapy vs Placebo in the Treatment of Adult Patients With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Oct 1;79(10):953-962. doi: 10.1001/jamapsychiatry.2022.2096. PMID 36001306
- [Background] Carhart-Harris RL, Bolstridge M, Day CMJ, Rucker J, Watts R, Erritzoe DE, Kaelen M, Giribaldi B, Bloomfield M, Pilling S, Rickard JA, Forbes B, Feilding A, Taylor D, Curran HV, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: six-month follow-up. Psychopharmacology (Berl). 2018 Feb;235(2):399-408. doi: 10.1007/s00213-017-4771-x. Epub 2017 Nov 8. PMID 29119217
- [Background] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667
- [Background] Goodwin GM, Aaronson ST, Alvarez O, Arden PC, Baker A, Bennett JC, Bird C, Blom RE, Brennan C, Brusch D, Burke L, Campbell-Coker K, Carhart-Harris R, Cattell J, Daniel A, DeBattista C, Dunlop BW, Eisen K, Feifel D, Forbes M, Haumann HM, Hellerstein DJ, Hoppe AI, Husain MI, Jelen LA, Kamphuis J, Kawasaki J, Kelly JR, Key RE, Kishon R, Knatz Peck S, Knight G, Koolen MHB, Lean M, Licht RW, Maples-Keller JL, Mars J, Marwood L, McElhiney MC, Miller TL, Mirow A, Mistry S, Mletzko-Crowe T, Modlin LN, Nielsen RE, Nielson EM, Offerhaus SR, O'Keane V, Palenicek T, Printz D, Rademaker MC, van Reemst A, Reinholdt F, Repantis D, Rucker J, Rudow S, Ruffell S, Rush AJ, Schoevers RA, Seynaeve M, Shao S, Soares JC, Somers M, Stansfield SC, Sterling D, Strockis A, Tsai J, Visser L, Wahba M, Williams S, Young AH, Ywema P, Zisook S, Malievskaia E. Single-Dose Psilocybin for a Treatment-Resistant Episode of Major Depression. N Engl J Med. 2022 Nov 3;387(18):1637-1648. doi: 10.1056/NEJMoa2206443. PMID 36322843